CLINICAL TRIAL: NCT01778101
Title: A Pilot Study - Lansoprazole in Preterm Infants With Gastroesophageal Reflux
Brief Title: Lansoprazole in Preterm Infants With Reflux
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han-Suk Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lanso_pilot; 0720120860 (Other Grant/Funding Number: Konect)
Record Dates: First submitted 2013-01-13; First posted 2013-01-29 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Preterm Infants; Gastrointestinal Reflux
Keywords: preterm infants; reflux; impedance; pH; monitoring; lansoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lansoprazole (Experimental): lansoprazole 1mg/kg twice a day for 14days
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — lansoprazole 1mg/kg twice a day for 14days
  Other Names: lanston LFDT

SUMMARY:
This study is pilot study to evaluate safety and efficacy of lansoprazole in preterm infants with gastroesophageal reflux documented by 24hr pH impedance monitoring

ELIGIBILITY:
Inclusion Criteria:

* preterm infant
* documented gastrointestinal reflux by 24hr pH monitoring

Exclusion Criteria:

* unstable vital sings
* congenital anomaly in upper gastrointestinal tract incuding esophagus
* drug history of H2 blocker during last 1 week
* medication of warfarin, carbamazepine, phenytoin, rifampin
* renal or hepatic dysfunction
* inappropriate clinical conditions judged by researchers

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
impedance pH monitoring | day14
  number of acid exposure percent time of acid exposure mean acid clearance time Acid Reflux Composite Score Analysis ; total time in reflux, episodes of 5min, composite score Bolus exposure(impedance); acid percent time, weakly acid percent time, weakly alkaline percentime Reflux Episodes activity Reflux Symptom Index Reflux Symptom Sensitivity Index Reflux Symptom Association Probability

SECONDARY OUTCOMES:
Symtomts of reflux_d5 | day 5
  apnea bradycardia desaturation regurgitate vomiting
impedance pH monitoring_d10 | day10
  number of acid exposure percent time of acid exposure mean acid clearance time Acid Reflux Composite Score Analysis ; total time in reflux, episodes of 5min, composite score Bolus exposure(impedance); acid percent time, weakly acid percent time, weakly alkaline percentime Reflux Episodes activity Reflux Symptom Index Reflux Symptom Sensitivity Index Reflux Symptom Association Probability
impedance pH monitoring_d5 | day5
  number of acid exposure percent time of acid exposure mean acid clearance time Acid Reflux Composite Score Analysis ; total time in reflux, episodes of 5min, composite score Bolus exposure(impedance); acid percent time, weakly acid percent time, weakly alkaline percentime Reflux Episodes activity Reflux Symptom Index Reflux Symptom Sensitivity Index Reflux Symptom Association Probability
Symtomts of reflux_d10 | day 10
  apnea bradycardia desaturation regurgitate vomiting
Symtomts of reflux_d14 | Symtomts of reflux_d14 day 14
  apnea bradycardia desaturation regurgitate vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Han-Suk Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Children's Hospital, Seoul, South Korea